CLINICAL TRIAL: NCT02525211
Title: Double-blind Randomized Prospective Phase III Study of a Continues Cicatricial Perfusion of Ropivacaine Versus Placebo After Mastectomy : Rehabilitation After Treatment of the Postoperative Pain From Hospital to Home
Brief Title: Continues Cicatricial Perfusion of Ropivacaine Versus Placebo After Mastectomy : Rehabilitation After Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment defect
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOLOSEIN / IPC 2011-005
Record Dates: First submitted 2012-11-16; First posted 2015-08-17 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine (Experimental): Ropivacaine
  Interventions: Drug: Ropivacaine
- placebo (Placebo Comparator): physiological saline
  Interventions: Drug: physiological saline

INTERVENTIONS:
Drug: Ropivacaine — a bolus of 10 ml of ropivacaine 7,5 mg / l then by a diffuser of local anesthesic (Ropivacaine 2mg / ml in continuous flow 10ml / hour) connected on the catheter the day after the intervention before returning at home
  Arms: Ropivacaine
Drug: physiological saline — a bolus of 10 ml of physiological saline in the catheter of multi- drilled cicatricial perfusion
  Arms: placebo

SUMMARY:
The acute pain care, in particular after breast cancer surgery must be early and quickly effective, because a severe postoperative pain increases the risk of chronic pain and exposes to a risk of important embarrassment for the realization of simple daily movements.

Associated to conventional analgesics administered by systemic way, a local anesthesic (ropivacaine) can be continuously infused (Continues Cicatricial Perfusion CCP) in the operating wound by a multi-drilled catheter by means of a elastomeric diffuser set up in the surgical unit by the surgeon at the end the surgical procedure.

Besides the control of the postoperative acute pain, the local anesthesic could intervene in the prevention of the chronic pain, the early recovery, the reduction of the neuropathic pains and the decrease of needs in morphine after mastectomy.

The duration of hospitalization being lower than 48 hours for this type of surgery, the investigators envisage an immediate follow-up in the Units of Care then at home, what will require a training of the hospital actors and at home (patient, family, visiting nurse, general practitioner).

Although proposed for several years, the CCP after breast surgery is still a little spread technique and few works had evaluated the pain at rest and at mobilization after mastectomy, the early rehabilitation, and to spread its use towards home, that is why we propose a randomized double-blind study ropivacaine / placebo in patients after mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years,
* Operated for a breast cancer by mastectomy with or without lymph node dissection, without immediate reconstruction,
* Capable of understanding the antalgic protocol,
* No contraindication to the local anesthesics,
* Social security affiliation,
* Signed informed consent.

Exclusion Criteria:

* Preoperative radiotherapy,
* Local infection,
* Contra-indication to the local anesthetic or to CCP,
* Contra-indication for the use of morphine,
* Contra-indication for the use of remifentanil,
* Addiction to opioid analgesics know or not,
* Allergy to local anesthetics,
* Hepatic or renal impairment grim known,
* Previous surgery on the operated breast,
* Pregnant women, or child-bearing potential, or lactating women,
* Patient deprived of liberty or under supervision of a guardian.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Delay to obtain the three criteria of premature recovery after mastectomy | time from surgery up to 6 months (At day of surgery, and at day 1, day 2, day 3 and day 15, then at month 3 and month 6).
  Delay to obtain the three criteria of premature recovery after mastectomy until 3 months post surgery:satisfactory analgesia defined by a Digital Scale lower than 4, estimated at rest and after standardized mobilization in immediate postoperative, and recourses or not to an analgesia of help, and capacity to drink with a glass and to thread the sleeve of a garment with the member side of the operated breast.

SECONDARY OUTCOMES:
pain intensity | time from surgery up to 6 months (At day of surgery, and at day 1, day 2, day 3 and day 15, then at month 3 and month 6).
  postoperative global and neuropathic pain scale
Analgesics consumption measure | time from surgery up to 3 months (At day of surgery, and at day 1, day 2, day 3 and day 15, then at month 3 and month 6).
  - Consumption of analgesics taken at request, in particular morphine savings in immediate postoperative
Measure of side effects rate | from surgery up to 3 days after the end of treatment
  - Side effects evaluated according to CTC-AE V4 (COMMON TERMILOLOGY CRITERIA FOR ADVERSE EVENTS version 4)
quality of life evaluation | time from surgery up to 3 months (At day of surgery, and at day 1, day 2, day 3 and day 15, then at month 1 and month 3).
  - Satisfaction and quality of life of the patients evaluated by scale and questionaries (QLQ-C30)at inclusion, month 1, month 3.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel FRANCON, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Daniel FRANCON, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr